CLINICAL TRIAL: NCT01920295
Title: Safety and Efficacy of Cryoballoon Ablation of Atrial Fibrillation as First-line Therapy
Acronym: C-frost
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuksek Ihtisas Hospital (Other)
Responsible Party: Principal Investigator, Serkan Cay, Associate Professor, Yuksek Ihtisas Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3196568
Record Dates: First submitted 2013-05-01; First posted 2013-08-09 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cryoballoon ablation (Experimental): Cryoballoon ablation
  Interventions: Device: Cryoballoon ablation
- Cryoballoon after medical therapy (Active Comparator): Cryoballoon ablation
  Interventions: Device: Cryoballoon ablation
- Cryoballoon as first-line therapy (Experimental): Cryoballoon ablation
  Interventions: Device: Cryoballoon ablation
- Cryoballoon after failed drug therapy (Active Comparator): Cryoballoon ablation
  Interventions: Device: Cryoballoon ablation

INTERVENTIONS:
Device: Cryoballoon ablation

SUMMARY:
Cryoballoon ablation of paroxysmal atrial fibrillation can be used as first-line therapy compared to second choice after failed medical therapy

ELIGIBILITY:
Inclusion Criteria:

* paroxysmal atrial fibrillation, symptomatic

Exclusion Criteria:

* atrial fibrillation other than PAF, asymptomatic, previous AF ablation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Recurrent atrial fibrillation, atrial flutter and atrial tachycardia (composite) | 12 months from the procedure
  At prespecified interval of 12th month from the index procedure occurence of Recurrent atrial fibrillation, atrial flutter and atrial tachycardia ( Number of Participants with Recurrent atrial fibrillation, atrial flutter and atrial tachycardia )was assessed using ambulatory holter ECG monitoring
Recurrent atrial fibrillation, atrial flutter and atrial tachycardia (composite) | 3 months from the procedure
  At prespecified interval of 3rd month from the index procedure occurence of Recurrent atrial fibrillation, atrial flutter and atrial tachycardia ( Number of Participants with Recurrent atrial fibrillation, atrial flutter and atrial tachycardia )was assessed using ambulatory holter ECG monitoring
Recurrent atrial fibrillation, atrial flutter and atrial tachycardia (composite) | 6 months from the procedure
  At prespecified interval of 6th month from the index procedure occurence of Recurrent atrial fibrillation, atrial flutter and atrial tachycardia ( Number of Participants with Recurrent atrial fibrillation, atrial flutter and atrial tachycardia )was assessed using ambulatory holter ECG monitoring
Recurrent atrial fibrillation, atrial flutter and atrial tachycardia (composite) | 9 months from the procedure
  At prespecified interval of 9th month from the index procedure occurence of Recurrent atrial fibrillation, atrial flutter and atrial tachycardia ( Number of Participants with Recurrent atrial fibrillation, atrial flutter and atrial tachycardia )was assessed using ambulatory holter ECG monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- Yuksek Ihtisas Heart-Education and Research Hospital, Ankara, Turkey (Türkiye)